CLINICAL TRIAL: NCT02413164
Title: Effectiveness of a Multimodal Physical Therapy Program on Clinical Symptomatology and Physical Fitness in Persons With Schizophrenia
Brief Title: Multimodal Physical Therapy Program in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD, University of Malaga
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12-2014
Record Dates: First submitted 2015-03-24; First posted 2015-04-09 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mental Health; Physical Therapy; Quality of life; Stigma; Positive and negative symptoms; Physical fitness; Physical activity
MeSH Terms: conditions — Schizophrenia; Psychological Well-Being; Social Stigma; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical intervention group (Experimental): 12 weeks of groupal sessions of individualised multimodal physiotherapy programme of therapeutic exercises with education healthy-style-of-life based, 2 times for week.
  Interventions: Other: A multimodal physiotherapy programme
- Control group (No Intervention): This group will receive usual care and will be in wait list status for the duration of study, later the intervention will be offered to this group.

INTERVENTIONS:
Other: A multimodal physiotherapy programme — Intervention: individualised Multimodal Physiotherapy Programme of therapeutic exercises with education healthy-style-of-life based.
  Groupal sessions two times per week during 12 weeks. Each session 60 minutes: 10 minutes of warm up, 20 minutes of strength and muscular endurance, 20 minuts of aerobic training, 10 minutes of cold-down.
  Intensity aerobic training: The training heart rate will be calculated according to recommendations of the American College of Sport Medicine (ACSM), it must oscillate between 55/65% and 90% of the HRmax. Initial four weeks: moderate intensity (55-69% HRmax); Following weeks according to each response, to higher level of training (70-89% HRmax). Strength training: individualised working with the principal muscular groups. 3 sessions using a weight which can repeat the exercise 10-15 times, increasing to a weight at which they can repeat the exercise 8-12 times.
  Arms: Physical intervention group

SUMMARY:
The aim of the investigators' study would evaluate the effectiveness of a multimodal exercise program on physical fitness, physical activity level and clinical symptomatology in patients with schizophrenia.

DESIGN: Randomized controlled trial. SUBJECTS OF THE STUDY: People with schizophrenia who receiving treatment in Regional Hospital of Malaga. INTERVENTION: DATA ANALYSIS: descriptive statistics, measuring central tendency and dispersion of the variables study. Inferential statistics will be made between intervention of key variables and outcome.

DETAILED DESCRIPTION:
It´s well known that life expectancy of people with severe mental disorders is approximately from 15 to 20 years less compared with general population. The higher mortality risk in this population group reflects a combination of factors: a) increased prevalence of comorbid medical conditions; b) adverse effects of pharmacological treatment; c) higher rates of suicide, accidental and other violent death; d) poorer access to physical healthcare than for the general population. In addition, this vulnerable population has an extremely high prevalence of obesity, nearly twice that of the overall population. Therefore, it is not surprising that persons with serious mental illness have an increased occurrence of weight-related conditions, including heightened risk of diabetes mellitus, hypertension, and dyslipidaemia; in addiction to this, these pathologies are under-diagnosed and under-treated. Environmental issues and unhealthy lifestyle can account for all these conditions, particularly in people with SMI, such as high levels of cigarette smoking, unhealthy diet or sedentary life style. Tendency to isolation and a reduced social network are often obstacles to the practice of physical exercise.

In addition, antipsychotics, in particular atypical antipsychotics, have been associated with weight gain, dyslipidaemia, diabetes, and other cardiac risk factors. Furthermore, the side effects of these medications are one of the most significant barriers to changing their lifestyle.

Finally, the stigma associated with mental illness may also contribute to low levels of participation in mainstream leisure-time physical activities.

Regular practise of physical exercise improves physical and mental health in the general population. A recent systematic review of physical activity and schizophrenia has shown improvement in both positive and negative symptoms, and a general increase in wellbeing of people with schizophrenia. In addition to cardiac and metabolic effects, physical exercise has demonstrated an improvement in both depression and anxiety.

The main objective of this study is to evaluate the effectiveness of a multimodal physical activity programme in physical fitness and physical activity level in persons with a diagnosis of schizophrenia.

Secondary objectives are: Evaluate the effect of this intervention in clinical symptomatology; Analyse the effect of this programme in motivating these persons to undertake physical activity; Identify the effect of the program on the physical fitness of the subjects; Evaluate any influence of the program on the self-perception of stigma in the subjects; Evaluate any variation of level of physical activity before and after the study in the subjects; Measure the impact on the quality of life of people who participate in this study; Perform a cost-effectiveness analysis of the program.

The present study is a randomized clinical trial to compare the effect of a multimodal, individualized, physical programme of muscular strength, endurance, aerobic training and health education against a control group.

All variables will be measured at the beginning and the end of the 12-week program by the same evaluator, whose group of subjects will be randomly allocated to the trial group and control group without their knowledge. Furthermore, the variables will be measured 9 months after the end of the program. Subjects allocated to the control group will have all the same variables measured, and will be given the option to participate in the program once the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Persons with diagnosis of schizophrenia
* Have agreed to agreeing to participate in the study
* Have signed the informed consent
* Be able to complete scales and perform physical tests

Exclusion Criteria:

* Have a contraindication for performing physical intervention.
* Destabilization of the symptoms
* Be participating in a program of structured physical activity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Baseline, 4 moth (Postintervention) and 13 month from baseline (9 months postintervention)
  The Positive and Negative Syndrome Scale--Spanish adaptation. Peralta V. Psychometric properties of the positive and negative syndrome scale (PANSS) in schizophrenia.
  The spanish version of this scale has a (CCI=0.71 for possitive symptoms; CCI=0.80 for negative symptoms; CCI=0.56 In General psycopatology).

SECONDARY OUTCOMES:
International Physical activity Questionnaire. Short form (IPAQ-7) | Baseline, 4 moth (Postintervention) and 13 month from baseline (9 months postintervention)
  The short version will be used centred on the time and intensity of the physical activity undertaken by the subject in the last 7 days.
Physical activity (accelerometry) | Baseline, 4 moth (Postintervention) and 13 month from baseline (9 months postintervention)
  For measure the physical activity level of participants an accelerometer will be use during 9 days (dismissing the first and the last days for analysis data)
Self-efficacy and social support for physical activity (SS/SE) | Baseline, 4 moth (Postintervention) and 13 month from baseline (9 months postintervention)
  Adaptation and psychometric properties of the self-efficacy/social support for activity for persons with intellectual disability scale (SE/SS-AID) in a Spanish sample.
12-Item Short-Form Health Survey | Baseline, 4 moth (Postintervention) and 13 month from baseline (9 months postintervention)
  Reliability and validity of the SF-12 health survey among people with severe mental illness.
Internalized Stigma of Mental Health questionnaire | Baseline, 4 moth (Postintervention) and 13 month from baseline (9 months postintervention)
  Internalized stigma of mental illness: psychometric properties of a new measure.
  Proposal of a socio-cognitive-behavioral structural equation model of internalized stigma in people with severe
Self-determination motivation in physical fitness | Baseline, 4 moth (Postintervention) and 13 month from baseline (9 months postintervention)
  self-determination motivation in a physical fitness setting: validation of the Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2) in a Spanish sample.
Client Service Receipt Inventory (CSRI). | Baseline, 4 moth (Postintervention) and 13 month from baseline (9 months postintervention)
  The cost effectiveness will be measured by evaluating the services used by the subjects using the Spanish version of the Client Service Receipt Inventory (CSRI).
  Client Socio-Demographic and Service Receipt Inventory-European Version: development of an instrument for international research. EPSILON Study 5. European Psychiatric Services: inputs Linked to Outcome Domains and Needs. Br J Psychiatry, Suppl. 2000;39:28-63 Vázquez-Barquero J, Gaite L, Cuesta M, García-Usieto E, Knapp M, Beecham J. Versión española del CSRI: una entrevista para la evaluación de costes en salud mental. Arch Neurobiol (Madr). 1997;60(2):171-84.
  This is a structured interview with either the subjector their carers, to obtain retrospective information about the use of health and social services in the past 12 months.
Physical fitness (6-min walk test, Timed up and go test, 30 seconds sit to stand test, handgrip test) | Baseline, 4 moth (Postintervention) and 13 month from baseline (9 months postintervention)
  The 6 minute test. A test of cardiorespiratory function which consists in measuring the maximum distance the subject can cover in 6 six minutes using a standard procedure.
  Timed up and go test. This is a test to evaluate mobility that requires both static and dynamic equilibrium. It measures the time that the subject takes to stand up from sitting, walk three metres, turn around and return to sit down in the seat.
  30 seconds sit to stand test(49,50). Measures the number of times that the subject can sit down in and stand up from a chair without using the support of the arms (arms will remain crossed across the chest during the test). This measures the strength of the legs.
  Handgrip test: This test is carried out using the recommendations of the American Association of Manual Therapies using a Jamar dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta Vargas, PhD, Principal Investigator — University of Malaga
Locations (1):
- IBIMA, Málaga, Málaga, Spain

REFERENCES:
- [Derived] Perez-Cruzado D, Cuesta-Vargas AI, Vera-Garcia E, Mayoral-Cleries F. The relationship between quality of life and physical fitness in people with severe mental illness. Health Qual Life Outcomes. 2018 May 2;16(1):82. doi: 10.1186/s12955-018-0909-8. PMID 29720196